CLINICAL TRIAL: NCT04972591
Title: Follow-up Study of Population Vaccinated With COVID-19 Vaccine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qin Ning (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Yichang Central People's Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Xiangya Hospital of Central South University (Other); Shiyan Renmin Hospital (Unknown); The second Hospital of JingZhou (Unknown); Yunnan Provincial Infectious Disease Hospital (Other); WUHAN NO.7 HOSPITAL (Unknown); Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ20210623
Record Dates: First submitted 2021-07-21; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: COVID-19; Vaccination; Anti-body
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cell (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CHB Group: Patients with CHB
- Compared Group: Healthy people

SUMMARY:
A multi-centered clinical follow-up study to investigate the long-term dynamic of COVID-19 antibody level after vaccination.

DETAILED DESCRIPTION:
From December 2019, coronavirus disease 2019 (COVID-19), caused by a β-coronavirus known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has spread across the globe. As of July 6, 2021, more than 180 million confirmed cases and around 4 million deaths have been reported globally. Till now, many treatment methods has gradually formed a consensus. At the same time, several domestic vaccines have been offered to the public for free inoculation in our country. However, due to the urgent form of the epidemic, the short vaccine development cycle and heavy tasks, there is no clear conclusion on the long-term changes in antibody levels after vaccination.Therefore, we plan to carry out a multi-center prospective observational trial to better understand the dynamic changes of the antibody levels in patients after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years old or elder) who prepare or have been vaccinated against COVID-19, and has not participated in similar clinical studies.

Exclusion Criteria:

* People who are allergic to any active ingredient of the vaccine, any inactive ingredient which was used in the production process, or those who have been allergic to the same kind of vaccine before.
* People who have had severe allergic reaction to vaccine before (such as acute allergic reaction, vascular neuroedema, dyspnea, etc.)
* People with uncontrolled epilepsy and other serious neurological diseases (such as transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.)
* People who are feverish, or suffering from acute diseases, or suffering from acute episodes of chronic diseases, or with serious chronic diseases without control.
* Pregnant woman
* Juvenile

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All population who has been vaccinated or are prepared to get vaccinated.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
symptoms and signs | 6months
  symptoms and signs after vaccination will be collected
antibody levels | 6months
  antibody levels will be collected
laboratory findings | 6months
  Clinical laboratory examination were obtained during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No